CLINICAL TRIAL: NCT03525002
Title: Dopamine Action on Metabolism Depending on Genetic Heterogeneity - a Randomized, Placebo-controlled Double Blind Study
Brief Title: Dopamine Action on Metabolism in Relation to Genotype
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: University Hospital of Cologne (Other); University Hospital Lübeck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DopamineGenetics01
Record Dates: First submitted 2018-05-02; First posted 2018-05-15 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Bromocriptine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- FTO SNP rs8050136 (AA), Placebo (Placebo Comparator): Participants with FTO SNP rs8050136 AA receiving matching Placebo
  Interventions: Other: Placebo
- FTO SNP rs8050136 (AA), Bromocriptine (Active Comparator): Participants with FTO SNP rs8050136 AAreceiving Bromocriptine up to 5 mg
  Interventions: Drug: Bromocriptine
- FTO SNP rs8050136 (CA), Placebo (Placebo Comparator): Participants with FTO SNP rs8050136 CA receiving matching Placebo
  Interventions: Other: Placebo
- FTO SNP rs8050136 (CA), Bromocriptine (Active Comparator): Participants with FTO SNP rs8050136 CA receiving Bromocriptine up to 5 mg
  Interventions: Drug: Bromocriptine
- FTO SNP rs8050136 (CC), Placebo (Placebo Comparator): Participants with FTO SNP rs8050136 CC receiving matching Placebo
  Interventions: Other: Placebo
- FTO SNP rs8050136 (CC), Bromocriptine (Active Comparator): Participants with FTO SNP rs8050136 CC receiving Bromocriptine up to 5 mg
  Interventions: Drug: Bromocriptine

INTERVENTIONS:
Drug: Bromocriptine — In each FTO genotype group participants will be randomly receive bromocriptine or placebo.
  Arms: FTO SNP rs8050136 (AA), Bromocriptine; FTO SNP rs8050136 (CA), Bromocriptine; FTO SNP rs8050136 (CC), Bromocriptine
Other: Placebo — In each FTO genotype group participants will be randomly receive bromocriptine or placebo.
  Arms: FTO SNP rs8050136 (AA), Placebo; FTO SNP rs8050136 (CA), Placebo; FTO SNP rs8050136 (CC), Placebo

SUMMARY:
Obesity is a widespread disease with increasing prevalence and associated with serious secondary complications. So far, the origin of the disease, regardless of an existing positive energy balance, is not fully understood. In addition to environmental factors, the genetic background plays an important role in the pathogenesis of obesity. Of common genetic polymorphisms, variants in the fat mass and obesity associated gene (FTO) locus have the highest effect size on body weight. Animal and first clinical studies indicate that FTO variants interact with dopamine signaling in the brain, thus influencing the risk of overweight. In fact, preliminary results indicate that enhancing dopamine signaling with the dopamine agonist bromocriptine, depending on the FTO genotype, either induces weight loss or has a neutral effect on body weight.

The planned clinical trial serves to develop a genotype-specific and thus individualized therapy approach for obesity. The influence of dopamine agonist therapy on weight loss as a function of the FTO (rs8050136) genotype is to be tested.

Here, the greatest weight loss is expected to occur in subjects carrying the homozygous risk-allele (AA).

So far, there are only a few established conservative therapy forms of obesity, so that bariatric interventions with an increasing rate are necessary to achieve weight loss and thus a reduction in overall morbidity and mortality. Among the approved drug therapies for obesity, bromocriptine is commonly used. In addition, some interventions require injections. An early, conservative individualized, genotype-specific treatment with little side-effects would enable simple treatment of obesity.

Study design: 150 obese (BMI > 30) subjects (50 / study center) will be enrolled in the study. The subjects will be stratified according to their FTO genotype (rs8050136). Subjects will be randomized into placebo or bromocriptine treatment group. Treatment will last for 18 weeks and a follow-up will be performed 30 weeks after baseline.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between >30 kg/m².
* Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures.
* Females of childbearing potential (FCBP) must agree to utilize a reliable form of contraception simultaneously or practice complete abstinence from heterosexual contact while participating in the study.
* Males must agree to use a latex condom during any heterosexual contact while participating in the study and to refrain from donating semen or sperm while participating in this study.

Exclusion Criteria:

* Women during pregnancy and lactation.
* History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal products.
* Participation in other clinical trials or observation period of competing trials up to 30 days prior to this study.
* Diabetes mellitus
* Treatment with Methyldopa, levodopa, dopamine agonists, metoclopramid, domperidon, glycerol nitrate, griseofulvin, azol-antimycotic drugs, macrolide-antibiotics, octreotide, orlistat, tamoxifen, liraglutide
* Any relevant cardiovascular disease, e.g. myocardial infarction, acute coronary syndrome, unstable angina pectoris, Percutaneous transluminal coronary angioplasty (PTCA), heart failure (NYHA III-IV), stroke or transient ischemic attack (TIA)
* Acute or chronic viral hepatitis or liver cirrhosis
* Impaired renal function, defined as estimated Glomerular Filtration Rate (eGFR) ≤ 60 ml/min (MDRD formula) as determined during screening.
* Medical history of cancer and/or treatment for cancer within the last 5 years.
* Claustrophobia
* Any other clinically significant major organ system disease at screening such as relevant gastrointestinal, neurologic, psychiatric, endocrine (i.e. pancreatic), hematologic, malignant, infection or other major systemic diseases making implementation of the protocol or interpretation of the study results difficult.
* Presence of any contraindication for the conduct of an MRI investigation, such as cardiac pacemakers, ferromagnetic haemostatic clips in the central nervous system, metallic splinters in the eye, ferromagnetic or electronically operated active devices like automatic cardioverter defibrillators, cochlear implants, insulin pumps and nerve stimulators, prosthetic heart valves etc.
* hyperthyroidism
* therapy refractary hypertension
* peripheral arterial disease
* Parkinson´s disease
* Known current presence or history of one of the following psychiatric diseases: depression, mania, anxiety and panic disorder, obsessive-compulsive disorder, schizophrenia, psychosis, addiction
* pituitary disease
* treatment with bromocriptine during 12 month before entering the trial
* dementia
* gastric or intestinal ulcer
* Persons with limited temperature sensation and / or elevated sensitivity to warming of the body
* Persons with a hearing disorder or a increased sensitivity for loud noises
* smoking
* Refusal to get informed of unexpected detected pathological findings

Any other clinical condition that would jeopardize subjects' safety while participating in this clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
Interaction between FTO genotype and treatment on change in body weight. | 18 weeks
  Interaction between FTO (single nucleotide peptide) SNP rs8050136 genotype and treatment (bromocriptine or placebo) on change in body weight.

SECONDARY OUTCOMES:
Effect of bromocriptine vs. placebo on body weight | 18 weeks
Effect of bromocriptine vs. placebo on dietary intake | 18 weeks
  Dietary intake will be monitored by food diaries
Effect of bromocriptine vs. placebo on processing of food cues in the brain | 18 weeks
  Processing of food cues in the brain will be assessed by functional magnetic resonance imaging before and after treatment with bromocriptine or placebo
Effect of bromocriptine vs. placebo on body fat distribution | 18 weeks
  Body fat distribution will be assessed by magnetic resonance imaging and magnetic resonance spectroscopy before and after treatment with bromocriptine or placebo
Effect of bromocriptine vs. placebo on whole body insulin sensitivity | 18 weeks
  Whole body insulin sensitivity will be quantified from 5 point 75g oral glucose tolerance test before and after treatment with bromocriptine or placebo
Effect of bromocriptine vs. placebo on insulin secretion | 18 weeks
  Insulin secretion will be quantified from 5 point 75g oral glucose tolerance test before and after treatment with bromocriptine or placebo
Effect of bromocriptine vs. placebo on glucose tolerance | 18 weeks
  Glucose tolerance will be assessed by 75g oral glucose tolerance test before and after treatment with bromocriptine or placebo
Effect of bromocriptine vs. placebo on brain insulin sensitivity | 18 weeks
  Brain insulin sensitivity will be assessed by functional magnetic resonance imaging combined with intranasal insulin administration before and after treatment with bromocriptine or placebo
Effect of bromocriptine vs. placebo on resting energy expenditure | 18 weeks
  Resting energy expenditure will be assessed by indirect calorimetry before and after treatment with bromocriptine or placebo
Effect of bromocriptine vs. placebo on physical activity | 18 weeks
  Physical activity will be monitored using an accelerometer
Effect of bromocriptine vs. placebo on serum prolactin concentrations | 18 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - University Hospital Cologne, Cologne
  - University Hospital Luebeck, Lübeck
  - University of Tuebingen, Department of Internal Medicine IV, Tübingen

IPD SHARING:
Plan to Share IPD: No